CLINICAL TRIAL: NCT02394600
Title: The Impact of Grass SLIT Treatment on Birch Pollen Induced Allergic Rhinitis - a Pilot Evaluation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Dr. Anne Ellis, Chair, Division of Allergy & Immunology, Queen's University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: EEU-MERCK 001
Record Dates: First submitted 2015-03-04; First posted 2015-03-20 (Estimated); Results first posted 2018-01-29 (Actual); Last update posted 2018-01-29 (Actual); Status verified 2017-06

CONDITIONS: Allergic Rhinoconjunctivitis
Keywords: rhinitis; allergy
MeSH Terms: conditions — Rhinitis; Hypersensitivity | interventions — Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Grastek® (Experimental): 48 participants will receive Grastek® once per day for 120 days. Grastek® is a standardized sublingual immunotherapy (SLIT) tablet containing 2800 BAU of standardized allergen extract from Timothy grass (Phleum pretense). This SLIT product is approved by Health Canada and the Food and Drug Administration (FDA) for the treatment of grass-pollen induced allergic rhinoconjunctivitis (AR) in Canada and the United States respectively.
  Interventions: Drug: Grastek®
- Placebo (Placebo Comparator): 48 participants will receive placebo once per day for 120 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Grastek® — one tablet daily for four months
  Arms: Grastek®
Drug: Placebo — one tablet daily for four months
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
This pilot study is a Phase IV, single center, placebo-controlled, parallel study design conducted using the Environmental Exposure Unit (EEU). The study will aim to be determine whether there are any benefits from Grastek® for the treatment of birch-pollen induced allergic rhinoconjunctivitis. Grastek® is a Health Canada and FDA approved sublingual immunotherapy (SLIT) for the treatment of grass-pollen induced allergic rhinoconjunctivitis. The EEU provides a closed environment in which participants are exposed to a predetermined, controlled, constant level of airborne pollen. 96 participants will complete this study and will either receive Grastek® or placebo in a 1:1 ratio. The study will consist of a screening visit, a pre-treatment pollen exposure visit, 60 days of treatment with Grastek® or placebo, two treatment visits and a follow-up pollen exposure visit.

ELIGIBILITY:
Inclusion Criteria:

1. Participant demonstrates understanding and has provided an appropriately signed and dated informed consent.
2. Male or Female, 18 to 65 years of age, at time of the Screening visit.
3. Participant has a history of at least moderate allergic rhinoconjunctivitis due to hypersensitivity to birch pollen for a minimum of 2 years.
4. Participant responds to the birch pollen and timothy grass pollen through a standard skin prick test administered at the Screening visit. A positive test will be defined as a wheal diameter at least 5mm or larger than the negative control (normal saline) wheal. A historical skin-prick test performed within three-hundred sixty-five (365) days or one (1) year at the site will be accepted in lieu of performing a new skin prick test.
5. Participant understands and is willing, able and likely to comply with study procedures and restrictions.
6. Participant, if female, has a negative urine pregnancy test at Visit 1 and is willing to use a medically acceptable form of birth control. Acceptable methods of birth control for this study include:

   * oral, patch, or intra-vaginal hormonal contraceptives
   * Norplant System®
   * Depo-Provera®
   * IUD
   * double barrier method
   * abstinence
   * surgically sterile females (hysterectomy or tubal ligation)
   * > 1 year post-menopausal females
   * same sex partner
   * partner vasectomy (> 3 months)
7. Participant is healthy as determined by pre-study medical history, physical examination and vital signs.
8. Participant is able to read, comprehend, and record all information in English.
9. Participant has a serum specific IgE level to both birch and timothy grass of ≥0.7 ku/L.

Exclusion Criteria:

1. Has significant current nasal or ocular symptoms that the study doctor associates with perennial allergic or non-allergic rhinitis.
2. Female participant who is pregnant or lactating.
3. Has a history of any illness that, in the opinion of the study investigator, might confound the results of the study or poses an additional risk to the participant by their participation in the study. This includes a clinically relevant medical or surgical history or presence of other respiratory disease (exceptions made for asthma and allergic rhinitis as defined in further exclusion criteria), or gastrointestinal, renal, hepatic, hematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, immunological, dermatological, connective tissue diseases or disorders, or a history of malignancy within the past 5 years, with the exception of non-melanoma skin cancer.
4. Has any significant abnormalities found during physical exam as determined by the investigator.
5. Has a current medical history of significant pulmonary disease and/or active asthma requiring daily drug therapy. Mild, intermittent asthma is permitted (managed with short acting beta-agonist less than 3 times per week). Isolated exercise-induced bronchospasm is also permitted.
6. Has received an investigational drug within the last thirty (30) days.
7. Has had use of immunotherapy containing grass or birch within the last 3 years.
8. Has significant nasal polyps, nasal septal perforation, or nasal tract malformations as noted on physical exam.
9. Administration of adrenaline (epinephrine) is contraindicated (e.g. participants with acute or chronic symptomatic coronary heart disease or concomitant beta-blocker therapy).
10. Is unlikely to cooperate with the requirements of the study including having the ability to communicate with the investigator appropriately.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2015-04; Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne K Ellis, MD, Principal Investigator — Queen's University
Locations (1):
- Kingston General Hospital, Kingston, Ontario, Canada

REFERENCES:
- [Derived] Ellis AK, Tenn MW, Steacy LM, Adams DE, Day AG, Walker TJ, Nolte H. Lack of effect of Timothy grass pollen sublingual immunotherapy tablet on birch pollen-induced allergic rhinoconjunctivitis in an environmental exposure unit. Ann Allergy Asthma Immunol. 2018 May;120(5):495-503.e2. doi: 10.1016/j.anai.2018.02.003. Epub 2018 Feb 9. PMID 29432967

RESULTS

PARTICIPANT FLOW:
Groups:
- Grastek: 4 months of once per day Grastek sublingual immunotherapy
- Placebo: 4 months of once per day matching placebo sublingual tablet
Period: Overall Study
Arm/Group | Grastek | Placebo
Started | 47 | 46
Completed | 43 | 44
Not Completed | 4 | 2
Not completed — Adverse Event | 3 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Grastek | Placebo | Total
Number analyzed (Participants) | 47 | 46 | 93
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 45 | 46 | 91
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Full Range); unit: years] | 37.89 [18 to 65] | 38.17 [22 to 58.75] | 38.03 [18 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 23 | 48
  Male | 22 | 23 | 45
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 47 | 46 | 93

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Nasal Symptom Score (TNSS) From Baseline to Post-treatment.
Description: To determine the effect of 4 months of treatment with Grastek® on the symptoms of birch pollen induced AR in participants with both timothy grass pollen-induced and birch pollen-induced allergen rhinitis (AR)
  TNSS is comprised of the sum of 4 symptoms: runny nose, itchy nose sneezing and nasal congestion. Each of these symptoms are evaluated based on a 4 point Likert scale from 0-3. 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms and 3 = severe symptoms. TNSS can therefore have a range from 0 to 12.
Time Frame: 4 months
Population: 93 participants were randomized into this study. The final number of participants that completed and were included for analysis are listed above.
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Groups:
- Placebo: 4 months of once per matching placebo sublingual tablet
Arm/Group | Grastek | Placebo
Number analyzed (Participants) | 43 | 44
Scores on a scale | 2.3 [1.5 to 3.1] | 2.2 [1.4 to 3.0]

2. Secondary Outcome: Analysis of Blood Samples for Potential Biomarkers by Comparing Baseline and Post-treatment Samples.
Description: To determine potential biomarkers predictive of clinical efficacy for birch pollen-induced AR following treatment with Grastek®
Time Frame: 4 months
Population: As the primary outcome showed that there was no significant difference between Grastek and placebo this outcome was not able to be completed.
Arm/Group | Grastek | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Grastek®: 4 months of once per day Grastek sublingual immunotherapy
Arm/Group | Grastek® | Placebo
Serious Adverse Events (participants affected / at risk) | 0/47 | 1/46
Other Adverse Events (participants affected / at risk) | 33/47 | 23/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Grastek® (N=47) | Placebo (N=46)
Worsening of ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Grastek® (N=47) | Placebo (N=46)
Upper respiratory tract infection (Infections and infestations) | 15 | 11
Nausea (Gastrointestinal disorders) | 4 | 2
Headache (General disorders) | 7 | 12
Ear pruritus (Ear and labyrinth disorders) | 8 | 0
Palate pruritus (General disorders) | 4 | 1
Sublingual pruritus (General disorders) | 7 | 0
Throat pruritus (General disorders) | 11 | 1
Tongue pruritus (General disorders) | 6 | 0
Nasal congestion (General disorders) | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No